CLINICAL TRIAL: NCT03107832
Title: Comparison of Bi-spectral Index-Controlled Sedation During a Thoracic Epidural Anesthesia With General Anesthesia in Laparoscopic Cholecystectomy
Brief Title: Thoracic Epidural Versus General Anaesthesia in Cholecystectomy
Acronym: EVGAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Murat Bilgi, associate professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbantIBU mb2
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- general anesthesia (Active Comparator): In general anesthesia group (Group G), and induction was managed using 1.5 mg/kg fentanyl and 2 mg/kg propofol; 0.5 mg/kg rocuronium and sevoflurane in a 50% oxygen /air mixture was used. Blood gas analysis monitoring was performed in the 30th minute before and after pneumoperitoneum
  Interventions: Procedure: thoracic epidural anesthesia procedure
- thoracic epidural anesthesia (Experimental): In epidural anesthesia group(Group E), a catheter was installed and received 20 mg lidocaine hydrochloride, 15 mg bupivacaine, and 25 mg fentanyl citrate adjusted to 10 cc with normal saline to be injected by the epidural catheter. Bi-spectral index -controlled sedation was provided
  Interventions: Procedure: thoracic epidural anesthesia procedure

INTERVENTIONS:
Procedure: thoracic epidural anesthesia procedure — general anesthesia procedure

SUMMARY:
CONTEXT AND AIMS: The aim of the study is to compare patients satisfaction of thoracic epidural and general anesthesia procedures in patients undergoing elective laparoscopic cholecystectomy. SETTINGS AND DESIGN: This comparative randomized study was conducted Abant Izzet Baysal University hospital between October 2012 and 2014.Forty-five patients who were under American Society of Anesthesiologists I-II classification and were scheduled for elective laparoscopic cholecystectomy were included in the study. SUBJECTS AND METHODS: All participant was separated, two group. In epidural anesthesia group(Group E), a catheter was installed and received 20 mg lidocaine hydrochloride, 15 mg bupivacaine, and 25 mg fentanyl citrate adjusted to 10 cc with normal saline to be injected by the epidural catheter. Bispectral index -controlled sedation was provided. In general anesthesia group(Group G), and induction was managed using 1.5 mg/kg fentanyl and 2 mg/kg propofol; 0.5 mg/kg rocuronium and sevoflurane in a 50% oxygen/air mixture was used. Blood gas analysis monitoring was performed in the 30th minute before and after pneumoperitoneum. Surgical satisfaction was recorded after pneumoperitoneum. After the operation, 75 mg diclofenac sodium was applied for patients with Numeric Rating Scale scores higher than 4. STATISTICAL ANALYSIS USED:Data analysis was performed using the Statistical Package for the Social Sciences version 18 software (SPSS, Chicago, IL, US). Descriptive variables, such as age, ASA classification, weight, height, mean arterial pressure (MAP), HR, and duration of surgery, are given as mean ± standard deviation, and an independent sample t-test (normal distribution) as well as a Mann-Whitney U test (not a normal distribution) were used for continuous variables. To compare the normal and abnormal distributions in the groups, simple t-test, and Wilcoxon test was used, respectively. The results were considered statistically significant at p-values <0.05.

DETAILED DESCRIPTION:
This comparative randomized study included 45 patients in this study following receiving institutional ethical committee approval (Clinical Ethical Committee of Abant Izzet Baysal University, Bolu, Turkey. Ethical Committee Number: 2012/234) and collecting informed consent. Pre-anesthetic evaluations were conducted in these patients who were between the ages of 18 and 75 and fell into American Society of Anesthesiologists (ASA) risk categories I-II who were scheduled for elective laparoscopic cholecystectomy. Exclusion criteria; patients with any of the following: allergies against any of the drugs to be used in the study, current pregnancy, severe cardiac, renal, and liver diseases, previous upper abdominal surgery, acute cholangitis, a body mass index >32 kg m2, contraindications for epidural anesthesia and elective surgery.

All the patients received preoperative evaluations, were informed about the study, provided their informed consent, and were informed about the method of anesthesia to be applied In this study, present a comparison of patients and surgical satisfaction and hemodynamic changes of patients for whom an elective laparoscopic cholecystectomy procedure was planned.

ELIGIBILITY:
* Inclusion Criteria:

  * American Society of Anesthesiologists I-II classification ,
  * Elective laparoscopic cholecystectomy ,
  * Ages of 18 and 75
* Exclusion Criteria:

  * allergies against any of the drugs to be used in the study,
  * current pregnancy,
  * severe cardiac, renal, and liver diseases,
  * previous upper abdominal surgery,
  * acute cholangitis,
  * a body mass index >32 kg m2,
  * contraindications for epidural anesthesia and elective surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12-30 (Actual); Primary Completion 2013-08-25 (Actual); Study Completion 2013-12-29 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | after postoperative 24 hour
  four level patient satisfaction scale

SECONDARY OUTCOMES:
mean arterial pressure | intaoperative 0, 5, 10, 15, 30, and 45 minutes
  physiological parameter
heart rate | intaoperative 0, 5, 10, 15, 30, and 45 minutes
  physiological parameter
Blood gas analysis | intaoperative 0 and 35 minutes
  physiological parameter
Hypotension | During the operation
  adverse effect, A decrease in the mean arterial pressure under 60 mm Hg was considered to hypotension
Bradycardia | During the operation
  adverse effect,A decrease of the Heart rate under 50 beats per minute was considered bradycardia
Nausea / vomiting | postoperative 24 hour
  adverse effect
Shoulder pain | intraoperative and postoperative 24 hour
  adverse effect
Sore throat | postoperative 24 hour
  adverse effect

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Medical School,, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No